CLINICAL TRIAL: NCT03124784
Title: Accuracy of Oxygen Saturation (SpO2) Noninvasive Pulse Oximeter Sensor (RD Disposable) Under Motion Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TR33143-000190A
Record Dates: First submitted 2017-04-14; First posted 2017-04-24 (Actual); Results first posted 2018-03-23 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-02

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- RD Disposable Sensors (Experimental): All subjects are enrolled into the test group and all subjects received the RD Disposable Sensors
  Interventions: Device: RD Disposable Sensors

INTERVENTIONS:
Device: RD Disposable Sensors — Noninvasive pulse oximeter sensor

SUMMARY:
In this study, the level of oxygen within the blood will be reduced in a controlled manner by reducing the concentration of oxygen the study volunteer breathes. The accuracy of a noninvasive pulse oximeter sensor under motion conditions will be assessed by comparison to the oxygen saturation measurements from a laboratory blood gas analyzer.

ELIGIBILITY:
Inclusion Criteria:

* Competent non-smoking adults
* Must weigh a minimum of 110 pounds and no more than 250 pounds unless subject is over 6 feet tall.
* Subjects must understand and consent to be in the study.
* American Society of Anesthesiology Class 1 (Healthy subjects without any systemic disease at all).
* Subjects with hemoglobin greater than or equal to 11 g/dL.

Exclusion Criteria:

* Subjects with polished, gel or acrylic nails.
* Subjects with damaged and/or finger nail deformities.
* Subjects who have had caffeine consumption the day of the study.
* Subjects who have taken pain medication 24 hours before the study.
* Subjects who have any systemic disease at all.
* Subjects who do not understand the study and the risks.
* Subjects who smoke.
* Subjects who use recreational drugs.
* Subjects who are pregnant or nursing.
* Subjects having either signs or history of peripheral ischemia.
* Subjects with open wounds, lacerations, inflamed tattoos or piercings, visible healing wounds.
* Subjects with psychiatric conditions or are on psychiatric medications.
* Subjects who have had invasive surgery within the past year- including but not limited to major dental surgery, gallbladder, heart, appendix, major fracture repairs (involving plates/ screws), jaw surgery, Urinary tract surgery, plastic surgery, major ears, nose throat (ENT) surgery, joint replacement or gynecological surgeries.
* Subjects who have had minor surgery or conditions in the past two months including but not limited to minor foot surgery (bunion), arthroscopic procedure, blood donation, plasma donation, skin biopsy/ procedures, root canal, fractures, eye surgery, and other minor procedures.
* Subjects that have been on antibiotics had congestion, head colds, flu, ear infection, chest congestion will have a 2 week waiting period from the time of finishing medications or must have no more symptoms.
* Subjects with claustrophobia, or anxiety.
* Subjects who have been in severe car accidents or a similar type of accidents will have a 12 month waiting period, from the time of the accident.
* Subjects who have had a concussion will have a 12 month waiting period, from the time of the concussion.
* Subjects with chronic unresolved asthma, lung disease and respiratory disease. Allergies to lidocaine, latex, adhesives, or plastic.
* Subjects with finger deformities or injuries (specific finger will not be used).
* Subjects with heart conditions, diabetes or hypertension.
* Subjects with resting heart rates greater than 85 beats per minute (BPM) or below 45 BPM
* Subjects who have given birth naturally will have 6 month waiting period. Subjects who had a pregnancy terminated, a miscarriage or had a c-section will have a 12 month waiting period.
* Others deemed ineligible by the clinical staff.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2017-01-20 (Actual); Study Completion 2017-01-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo Corporation, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RD Disposable Sensors
Started | 27
Completed | 25
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Computer/Equip Malfunction | 1

BASELINE CHARACTERISTICS:
Arm/Group | RD Disposable Sensors
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 7
  Asian or Pacific Islander | 4
  Caucasian | 7
  Hispanic | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: SpO2 ARMS of Sensor Under Motion Conditions
Description: Accuracy will be determined by comparing the noninvasive blood oxygen saturation measurement of the pulse oximeter to that obtained from a blood sample and calculating the arithmetic root mean square error (Arms) value. In order to obtain the Arms value, the blood oxygen saturation measurement is subtracted from the pulse oximeter oxygen saturation measurement for a number of samples, the average of this difference is computed as the bias. The standard deviation of the differences is computed as the precision. The square root of the sum of the squares of bias and precision is computed as the Arms Error value.
Time Frame: 1-5 hours
Population: 2 subjects were excluded from data analysis: one due to adverse event and the other due to equipment malfunction.
Measure: Number; unit: % of oxygen saturated hemoglobin
Arm/Group | RD Disposable Sensors
Number analyzed (Participants) | 25
% of oxygen saturated hemoglobin | 1.31
Statistical Analysis 1: Comparison: RD Disposable Sensors; Accuracy Root Mean Square (ARMS); Test type: Equivalence — ARMS<= 3 %SpO2 Error per International Organization For Standardization (ISO) -80601-2-61 Pilot study Monte Carlo simulation provided 80% Power with 25 subjects for an expected ARMS< 3 % SpO2; ARMS = 0; Per ISO-80601-2-61, the Root Mean Square difference (SpO2-SaO2) is the measure of merit for desaturation studies

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the course of the study (within 1 month).
Arm/Group | RD Disposable Sensors
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 2/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RD Disposable Sensors (N=27)
Sensitivity at site of arterial line placement (Injury, poisoning and procedural complications) | 1 (1)
Irregular heart rate (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-22): https://cdn.clinicaltrials.gov/large-docs/84/NCT03124784/Prot_SAP_000.pdf